CLINICAL TRIAL: NCT04584840
Title: Conservative Versus Surgical Treatment for Medication Related Osteonecrosis of the Jaws (MRONJ) Stages I and II, a Quasi-experimental Clinical Trial With Discovery of Salivary Biomarkers
Brief Title: Initial Management of MRONJ Stages I and II, a Clinical Trial With Detection of Salivary Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Principal Investigator, Juan Martin Zarate Gonzalez, Principal Investigator, Fundació d'investigació Sanitària de les Illes Balears
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CI-202-17
Record Dates: First submitted 2020-09-28; First posted 2020-10-14 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Osteonecrosis of the Jaw, Bisphosphonate Induced; Osteonecrosis of the Jaw, Bisphosphonate Related
Keywords: Mronj; Dronj; Biomarkers; Saliva; Surgical treatment; Bronj
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Unicentric quasi-experimental clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (non-surgical treatment) (No Intervention): * Soft diet.
  * Suspension of the use of prostheses or intraoral devices.
  * Oral hygiene guidelines.
  * Topical antiseptics: in the form of mouthrinses with 0.12% chlorhexidine after every meal and clorhexidine gel over the exposed bone or fistula.
  * Systemic antibiotics: for patients in stage 2 in which active acute infection is detected with Amoxicillin/Clavulanic Acid 875/125 mg every 8 hours for 2 weeks. Those allergic to penicillin will receive clindamycin 300 mg every 8 hours for 2 weeks or Levofloxacin 500 mg / day for 2 weeks. Systemic antibiotic treatment can be prolonged indefinitely until infection and symptoms are controlled.
- Group 2 (surgical treatment) (Experimental): Same guidelines of conservative treatment plus surgical treatment according to the following protocol:
  Specific protocol for surgical treatment:
  * Wide mucoperiosteal flaps and complete surgical excision of necrotic bone together with a mucosa margin of at least 2 mm.
  * Removal of dental pieces included in the diseased area and regularization of bony margins avoiding leaving sharp edges or spicules.
  * Secure a two layered waterproof closure without tension (simple or with local flaps).
  * Samples will be sent for Pathological and microbiological analysis.
  * Stitches removal after two weeks
  * Postoperative systemic antibiotic following the mentioned protocol until stitches removal.
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Same guidelines as group 1 (non-surgical) plus surgical treatment according to the following protocol:
  Specific protocol for surgical treatment
  * Wide mucoperiosteal flaps and complete surgical excision of necrotic bone together with a mucosa margin of at least 2 mm.
  * Removal of dental pieces included in the diseased area and regularization of bony margins avoiding leaving sharp edges or spicules.
  * Secure a two layered waterproof closure without tension (simple or with local flaps).
  * Samples will be sent for Pathological and microbiological analysis.
  * Stitches removal after two weeks
  * Postoperative systemic antibiotic following the mentioned protocol until stitches removal.
  Arms: Group 2 (surgical treatment)

SUMMARY:
Medication-related osteonecrosis of the jaw (MRONJ) is a serious complication in patients receiving antiresorptive therapies, such as Bisphosphonates and Denosumab. It is defined by the presence of exposed bone or a fistula that probes bone in the jaws for a period greater than 8 weeks in patient with a history of current or past antiresorptive or antiangiogenic treatment, and in the absence of prior radiotherapy or maxillary bone metastases. Depending on the severity of the disease 4 stages are described.

On the other hand, although the presence of alterations in the levels of certain biomarkers in saliva has been documented in patients with MRONJ compared to healthy patients, its applicability in clinical practice is still unknown.

Until recently, the status quo favored the adoption of a conservative strategy (non-surgical) for the initial management of patients with stage I and II. However, in recent years, this paradigm has been challenged by multiple authors who report better and more predictable outcomes with surgical treatment.

Based on the hypothesis that patients with MRONJ stage I and II subjected to initial surgical treatment have better results than those undergoing conservative (non-surgical) treatment, te research group has designed a unicentric, quasi-experimental clinical trial where the clinical and radiological outcome at the third month of 2 groups of patients with stages I and II MRONJ undergoing non-surgical treatment (Group 1 / control) versus initial surgical treatment (Group 2 / intervention) will be compared.

Also, the investigators hypothesize that the patients with complete resolution of the disease will also normalize salivary biomarkers levels unlike those with stable or progressive disease, meaning there is a correlation between clinical and biochemical response. Accordingly, the levels of specific salivary biomarkers at baseline and at the third month will be determined and compared with the clinical outcome.

After enrollment patients will be instructed and offered both treatment strategies, and assigned to the corresponding group according to their choice. Patients in group 1 (non-surgical) will receive traditional conservative treatment while patients undergoing surgical treatment will receive the same guidelines of conservative treatment plus surgery according to a specific surgical protocol.

DETAILED DESCRIPTION:
1. Type of study: unicentric quasi-experimental clinical trial
2. Hypothesis:

   2.1. Patients with MRONJ stage I and II subjected to initial surgical treatment have better results than those undergoing conservative (non-surgical) treatment.

   2.2. There is a correlation between clinical and biochemical outcome and the detection in saliva of certain biomarkers such as Amino Terminal Crosslinked Telopeptides of Type 1 Collagen (NTX), Matrix metallopeptidase 9 (MMP-9), Interleukin 1a (IL-1a), Interleukin 1b (IL-1b), Interleukin 6 (IL-6), Interleukin 17 (IL-17) and Interleukin 36α (IL-36α) may be useful to monitor treatment response.
3. Main Objectives:

   3.1. To compare the clinical and radiological outcome after 3 months of conservative treatment versus initial surgical treatment in patients with MRONJ stage I and II.

   3.2. To determine the levels of salivary biomarkers at the beginning and after 3 months of treatment while correlating them with the clinical outcome.
4. Secondary Aims

   * To determine if there is a relationship between the initial surface of exposed bone and the outcome.
   * To determine if clinical and radiological concordance in the outcome at the third month for each group.
   * To determine the rate of postoperative complications in the surgical group.
   * To determine if there is a relationship between the number of surgical interventions and the outcome.
   * To determine the percentage of patients undergoing conservative treatment which eventually end up requiring surgical treatment due to disease progression.
   * To determine the elapsed time until complete healing for both groups.
   * To determine the variables associated with a higher cure rate.
   * To determine the variables associated with increased risk of disease progression or recurrence.
5. MATERIAL AND METHODS 5.1. Sample Size Accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 21 patients per group are required to detect a cure rate of 30% and 70% in the conservative and surgical treatment group, respectively. Adding 10% to cover possible experimental losses, the sample increases to 23 per group.

5.2. Main Variables

* MRONJ Stage (1. Stage 1; 2. Stage 2).
* Type of treatment (GROUP 1/Control: Conservative Treatment, GROUP 2: Surgical Treatment).
* Clinical outcome at the third month
* Radiological outcome at the third month
* Levels of biomarkers in saliva at baseline and at the third month (NTX, MMP-9, IL-1a, IL-1b, IL-6, IL-17 and IL-36α). In the case scientific evidence of other relevant markers appears during the course of the study they may be included in the study.

5.3. Secondary Variables 5.3.1. Both groups

* Age (years)
* Sex (1.Man; 2.Mother)
* Diabetes (1. Yes; 2. No)
* Medication associated with the disease (1. Oral bisphosphonates, 2. Intravenous Bisphosphonates, 3. Denosumab, 4: Antiangiogenic).
* Underlying disease for antiresorptive therapy (1. Osteoporosis, 2. Cancer)
* Duration of treatment with medication associated with the disease.
* Factor that triggers the disease (1. Tooth Extraction; 2. Use of removable prosthesis; 3. Unclear cause)
* Suspension of medication associated with the development of MRONJ (1. Yes, 2. No)
* Concomitant treatment with corticosteroids (1. Yes, 2. No)
* Concomitant treatment with antiangiogenic drugs (1. Yes, 2. No)
* Visual Analogue Scale (VAS) pain in the inclusion visit, and in all follow-up visits.
* Exposed bone surface (1. mild: <0,5cm2; 2. Moderate: 0,5-2cm2; Severe:> 2cm2) or number of intraoral fistulas otherwise.
* Dimension of greater diameter of radiolucent area or sequestrum in the CT or Cone Beam-CT scan (cm)
* Time elapsed until complete healing.
* Recurrence.

5.3.2. Group 1 (Conservative medical treatment)

* Need for surgical treatment due to disease progression
* Time elapsed until surgical rescue treatment due to disease progression.

5.3.3. Group 2 (Surgical treatment)

* Postoperative complications.
* Number of interventions.

5.4. Inclusion Visit

* Patients will be informed about the different aspects of the study and will be given the information sheet to read carefully. Informed consent document will be given to read and sign.
* A thorough medical history will be collected including data about their socio-family environment, psychiatric illnesses and addictions.
* Complete and careful physical examination of the head and neck area will be carried out, including the measurement of the area of exposed bone in cm2 or, otherwise, the number of fistulas. Based on the clinical findings, stage 1 or 2 will be assigned according to the AAOMS guidelines.
* Once verified that the patient meets the inclusion criteria, patients will be assigned to the corresponding group according to their chosen treatment strategy.
* Radiological assessment will be carried out with Orthopantomography and CT-scan/Cone Beam-CT in all patients.
* Both groups will receive the same standard conservative treatment according to our protocol, meaning group 1 (non-surgical) will serve as control group.
* For patients enrolled in the surgical group, routine preoperative exams will be requested and surgical intervention will be scheduled within a maximum period of 3 weeks from the inclusion visit following a rigorous and standardized surgical protocol.

5.4.1 STANDARD PROTOCOL FOR CONSERVATIVE TREATMENT (applicable to both groups)

* Soft diet.
* Suspension of the use of prostheses or intraoral devices.
* Oral hygiene guidelines.
* Topical antiseptics: in the form of mouthrinses with 0.12% chlorhexidine after every meal and clorhexidine gel over the exposed bone or fistula.
* Systemic antibiotics: for patients in stage 2 in which active acute infection is detected with Amoxicillin/Clavulanic Acid 875/125 mg every 8 hours for 2 weeks. Those allergic to penicillin will receive clindamycin 300 mg every 8 hours for 2 weeks or Levofloxacin 500 mg / day for 2 weeks. Systemic antibiotics treatment can be prolonged indefinitely until infection and symptoms are controlled.

5.4.2. SPECIFIC PROTOCOL FOR SURGICAL TREATMENT

* Wide mucoperiosteal flaps and complete surgical excision of necrotic bone together with a mucosa margin of at least 2 mm.
* Removal of dental pieces included in the diseased area and regularization of bony margins avoiding leaving sharp edges or spicules.
* Secure a two layered waterproof closure without tension (simple or with local flaps).
* Samples will be sent for Pathological and microbiological analysis.
* Stitches removal after two weeks
* Postoperative systemic antibiotic following the mentioned protocol until stitches removal.

5.4.3. SALIVA COLLECTION PROTOCOL

* Patients must avoid rinsing and ingestion of solids or liquids for at least 1 hour prior to collection.
* The collection will take place between 8 and 10 am.
* Five minutes after an oral rinse with distilled water, 5 ml of unstimulated full saliva from the lower lip will be collected.
* The samples will be processed within the first hour of collection of the sample by centrifuging at 2,600 x g for 15 minutes at 4 ° C. The supernatant will be collected and stored at -80 ° C until the biomarkers are analyzed.

5.4.4. SUCCESSIVE VISITS

* Controls will be carried out 2 weeks after the inclusion visit and then monthly until the third month when the outcomes will be determined and the second sample of saliva will be collected. Long term follow-up will continue every three to six months depending on patient characteristics and desires.
* At each visit, the following information will be recorded: symptoms with VAS for pain; physical examination of head and neck; presence of exposed bone and surface in cm2 or number of fistulas otherwise. If complete mucosal healing is found, the time elapsed since the start of treatment will be recorded.
* Patients in GROUP 1, may develop disease progression refractory to conservative management. In that case, the second saliva sample will be collected before the third month and previous to surgical treatment.
* Patients of GROUP 2 with persistent disease, recurrence or significant worsening will undergo revision surgery if accepted.
* Radiological follow-up will be carried out with orthopantomography and CT scan/Cone Beam-CT at the third month.

5.4.5. STATISTICAL ANALYSIS Normality tests and graphs will be used to determine if the variables follow a normal distribution. Variables with normal distribution are expressed as mean ± standard deviation and those without normal distribution are expressed as median and interquartile range. To evaluate the differences between groups, the student's t test or the Mann-Whitney U test will be used for quantitative variables; and the chi-square test or Fisher's exact test for qualitative variables.

The correlations will be examined by the Spearman or Pearson rank correlation. Paired or related sample tests will be used to assess intragroup differences. A value of p <0.05 will be considered an indicator of a significant difference.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of stage I or stage II medication related osteonecrosis of the jaws (MRONJ) according to the 2014 AAOMS position paper.

Exclusion Criteria:

* Coexistence of any medical or social condition that prevents proper adherence to treatment or follow-ups (dependent patients without adequate socio-familiar support, drug addiction, severe psychiatric illness, terminal disease with life expectancy less than 3 months).
* Coexistence of Brown's Tumor, Paget's Disease or other bone diseases with the exception of Osteoporosis or bone metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Complete clinical resolution | Third month
  This is the first of the three possible clinical outcome. The patient has achieved complete mucosal healing meaning there is no signs of bone exposure or fistula, the patient is asymptomatic and thus, can be considered cured.
Clinically stable disease | Third month
  Second possible clinical outcome. The patient has not been cured but has neither gotten worse meaning that the area of bone exposure (in square centimeters) is equal or not greater than 50 percent of the initial measurement, and has not developed disease up-staging.
Clinical progression or up-staging | Third month
  Third possible clinical outcome. The patient has gotten worse meaning that the area of bone exposure (in square centimeters) is greater than 50 percent of the initial measurement, or the patient has progressed to a higher stage.
Level of salivary NTX | Third Month
  Expressed in nanomoles of bone collagen equivalents
Level of salivary MMP-9 | Third Month
  Expressed in nanograms/milliliters
Levels of IL-1a, IL-1b, IL-6, IL-17 and IL-36α. | Third Month
  Expressed in picograms/milliliters

SECONDARY OUTCOMES:
Radiological absence of radiolucent areas or complete ossification. | Third month
  This is the first of three possible radiological outcomes and means that the patient has no longer radiological signs of necrotic bone (sequestrum or osteolysis) in the CT or CB-CT scan.
Radiologically stable disease | Third Month
  Second possible radiological outcome. The radiolucent lesion or sequestrum (measured in centimeters by the greater diameter in the CT or CB-CT scan) is equal or not greater than 50 percent of the initial measurement, and does not meet radiological up-staging criteria.
Radiological progression | Third month
  Third possible radiological outcome. The radiolucent lesion or sequestrum (measured in centimeters by the greater diameter in the CT or CB-CT scan) is greater than 50 percent of the initial measurement, or meets radiological up-staging criteria.

CONTACTS AND LOCATIONS:
Overall Officials: MARTA MONJO CABRER, PHD, Study Director — Fundació d'investigació Sanitària de les Illes Balears; JOANA RAMIS MOREY, PHD, Study Director — Fundació d'investigació Sanitària de les Illes Balears; VICTOR A LASA MENÉNDEZ, MD, Study Chair; JUAN M ZÁRATE GONZÁLEZ, MD, Principal Investigator — Fundació d'investigació Sanitària de les Illes Balears
Locations (1):
- Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: IPD sharing subjected to prior authorization of the research group

REFERENCES:
- [Background] Ruggiero SL, Dodson TB, Fantasia J, Goodday R, Aghaloo T, Mehrotra B, O'Ryan F; American Association of Oral and Maxillofacial Surgeons. American Association of Oral and Maxillofacial Surgeons position paper on medication-related osteonecrosis of the jaw--2014 update. J Oral Maxillofac Surg. 2014 Oct;72(10):1938-56. doi: 10.1016/j.joms.2014.04.031. Epub 2014 May 5. PMID 25234529
- [Background] Bedogni A, Fusco V, Agrillo A, Campisi G. Learning from experience. Proposal of a refined definition and staging system for bisphosphonate-related osteonecrosis of the jaw (BRONJ). Oral Dis. 2012 Sep;18(6):621-3. doi: 10.1111/j.1601-0825.2012.01903.x. Epub 2012 Feb 22. No abstract available. PMID 22353421
- [Background] Schiodt M, Reibel J, Oturai P, Kofod T. Comparison of nonexposed and exposed bisphosphonate-induced osteonecrosis of the jaws: a retrospective analysis from the Copenhagen cohort and a proposal for an updated classification system. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Feb;117(2):204-13. doi: 10.1016/j.oooo.2013.10.010. Epub 2013 Nov 15. PMID 24332520
- [Background] Kolokythas A, Karras M, Collins E, Flick W, Miloro M, Adami G. Salivary Biomarkers Associated With Bone Deterioration in Patients With Medication-Related Osteonecrosis of the Jaws. J Oral Maxillofac Surg. 2015 Sep;73(9):1741-7. doi: 10.1016/j.joms.2015.03.034. Epub 2015 Mar 19. PMID 25889372
- [Background] Thumbigere-Math V, Michalowicz BS, de Jong EP, Griffin TJ, Basi DL, Hughes PJ, Tsai ML, Swenson KK, Rockwell L, Gopalakrishnan R. Salivary proteomics in bisphosphonate-related osteonecrosis of the jaw. Oral Dis. 2015 Jan;21(1):46-56. doi: 10.1111/odi.12204. Epub 2013 Nov 29. PMID 24286378
- [Background] Bagan J, Sheth CC, Soria JM, Margaix M, Bagan L. Bisphosphonates-related osteonecrosis of the jaws: a preliminary study of salivary interleukins. J Oral Pathol Med. 2013 May;42(5):405-8. doi: 10.1111/jop.12021. Epub 2012 Nov 15. PMID 23157469
- [Background] Bagan J, Saez GT, Tormos MC, Hens E, Terol MJ, Bagan L, Diaz-Fernandez JM, Lluch A, Camps C. Interleukin-6 concentration changes in plasma and saliva in bisphosphonate-related osteonecrosis of the jaws. Oral Dis. 2014 Jul;20(5):446-52. doi: 10.1111/odi.12150. Epub 2013 Jul 10. PMID 23837828
- [Background] Zhang Q, Atsuta I, Liu S, Chen C, Shi S, Shi S, Le AD. IL-17-mediated M1/M2 macrophage alteration contributes to pathogenesis of bisphosphonate-related osteonecrosis of the jaws. Clin Cancer Res. 2013 Jun 15;19(12):3176-88. doi: 10.1158/1078-0432.CCR-13-0042. Epub 2013 Apr 24. PMID 23616636
- [Background] Kim S, Williams DW, Lee C, Kim T, Arai A, Shi S, Li X, Shin KH, Kang MK, Park NH, Kim RH. IL-36 Induces Bisphosphonate-Related Osteonecrosis of the Jaw-Like Lesions in Mice by Inhibiting TGF-beta-Mediated Collagen Expression. J Bone Miner Res. 2017 Feb;32(2):309-318. doi: 10.1002/jbmr.2985. Epub 2016 Oct 12. PMID 27567012
- [Background] Bedogni A, Fedele S, Bedogni G, Scoletta M, Favia G, Colella G, Agrillo A, Bettini G, Di Fede O, Oteri G, Fusco V, Gabriele M, Ottolenghi L, Valsecchi S, Porter S, Petruzzi M, Arduino P, D'Amato S, Ungari C, Fung Polly PL, Saia G, Campisi G. Staging of osteonecrosis of the jaw requires computed tomography for accurate definition of the extent of bony disease. Br J Oral Maxillofac Surg. 2014 Sep;52(7):603-8. doi: 10.1016/j.bjoms.2014.04.009. Epub 2014 May 22. PMID 24856927
- [Background] Van den Wyngaert T, Claeys T, Huizing MT, Vermorken JB, Fossion E. Initial experience with conservative treatment in cancer patients with osteonecrosis of the jaw (ONJ) and predictors of outcome. Ann Oncol. 2009 Feb;20(2):331-6. doi: 10.1093/annonc/mdn630. Epub 2008 Oct 26. PMID 18953067
- [Background] Lerman MA, Xie W, Treister NS, Richardson PG, Weller EA, Woo SB. Conservative management of bisphosphonate-related osteonecrosis of the jaws: staging and treatment outcomes. Oral Oncol. 2013 Sep;49(9):977-983. doi: 10.1016/j.oraloncology.2013.05.012. Epub 2013 Jul 3. PMID 23830962
- [Background] Norholt SE, Hartlev J. Surgical treatment of osteonecrosis of the jaw with the use of platelet-rich fibrin: a prospective study of 15 patients. Int J Oral Maxillofac Surg. 2016 Oct;45(10):1256-60. doi: 10.1016/j.ijom.2016.04.010. Epub 2016 May 11. PMID 27179556
- [Background] Mucke T, Koschinski J, Deppe H, Wagenpfeil S, Pautke C, Mitchell DA, Wolff KD, Holzle F. Outcome of treatment and parameters influencing recurrence in patients with bisphosphonate-related osteonecrosis of the jaws. J Cancer Res Clin Oncol. 2011 May;137(5):907-13. doi: 10.1007/s00432-010-0953-1. Epub 2010 Oct 7. PMID 20927569
- [Background] Lesclous P, Grabar S, Abi Najm S, Carrel JP, Lombardi T, Saffar JL, Samson J. Relevance of surgical management of patients affected by bisphosphonate-associated osteonecrosis of the jaws. A prospective clinical and radiological study. Clin Oral Investig. 2014;18(2):391-9. doi: 10.1007/s00784-013-0979-2. Epub 2013 Apr 19. PMID 23604698
- [Background] Ruggiero SL, Kohn N. Disease Stage and Mode of Therapy Are Important Determinants of Treatment Outcomes for Medication-Related Osteonecrosis of the Jaw. J Oral Maxillofac Surg. 2015 Dec;73(12 Suppl):S94-S100. doi: 10.1016/j.joms.2015.09.024. PMID 26608159
- [Background] Carlson ER. Management of antiresorptive osteonecrosis of the jaws with primary surgical resection. J Oral Maxillofac Surg. 2014 Apr;72(4):655-7. doi: 10.1016/j.joms.2013.12.007. Epub 2013 Dec 15. No abstract available. PMID 24480762
- [Background] El-Rabbany M, Sgro A, Lam DK, Shah PS, Azarpazhooh A. Effectiveness of treatments for medication-related osteonecrosis of the jaw: A systematic review and meta-analysis. J Am Dent Assoc. 2017 Aug;148(8):584-594.e2. doi: 10.1016/j.adaj.2017.04.002. Epub 2017 May 18. PMID 28527518
- [Background] Hayashida S, Soutome S, Yanamoto S, Fujita S, Hasegawa T, Komori T, Kojima Y, Miyamoto H, Shibuya Y, Ueda N, Kirita T, Nakahara H, Shinohara M, Umeda M. Evaluation of the Treatment Strategies for Medication-Related Osteonecrosis of the Jaws (MRONJ) and the Factors Affecting Treatment Outcome: A Multicenter Retrospective Study with Propensity Score Matching Analysis. J Bone Miner Res. 2017 Oct;32(10):2022-2029. doi: 10.1002/jbmr.3191. Epub 2017 Jul 11. PMID 28585700
- [Background] Marx RE. Pamidronate (Aredia) and zoledronate (Zometa) induced avascular necrosis of the jaws: a growing epidemic. J Oral Maxillofac Surg. 2003 Sep;61(9):1115-7. doi: 10.1016/s0278-2391(03)00720-1. No abstract available. PMID 12966493
- [Background] Japanese Allied Committee on Osteonecrosis of the Jaw; Yoneda T, Hagino H, Sugimoto T, Ohta H, Takahashi S, Soen S, Taguchi A, Nagata T, Urade M, Shibahara T, Toyosawa S. Antiresorptive agent-related osteonecrosis of the jaw: Position Paper 2017 of the Japanese Allied Committee on Osteonecrosis of the Jaw. J Bone Miner Metab. 2017 Jan;35(1):6-19. doi: 10.1007/s00774-016-0810-7. Epub 2016 Dec 29. PMID 28035494
- [Background] Ristow O, Ruckschloss T, Muller M, Berger M, Kargus S, Pautke C, Engel M, Hoffmann J, Freudlsperger C. Is the conservative non-surgical management of medication-related osteonecrosis of the jaw an appropriate treatment option for early stages? A long-term single-center cohort study. J Craniomaxillofac Surg. 2019 Mar;47(3):491-499. doi: 10.1016/j.jcms.2018.12.014. Epub 2018 Dec 29. PMID 30642734
- [Background] Ristow O, Otto S, Troeltzsch M, Hohlweg-Majert B, Pautke C. Treatment perspectives for medication-related osteonecrosis of the jaw (MRONJ). J Craniomaxillofac Surg. 2015 Mar;43(2):290-3. doi: 10.1016/j.jcms.2014.11.014. Epub 2014 Nov 22. PMID 25541255